CLINICAL TRIAL: NCT00195299
Title: An Exploratory Biomarker Trail of Temsirolimus in Subjects With Newly Diagnosed Advanced Stage Squamous Cell Carcinoma of the Head & Neck
Brief Title: Study Evaluating Temsirolimus in Advanced Stage Squamous Cell Carcinoma of the Head & Neck
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 3066K1-147
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Squamous Cell Carcinoma
Keywords: Carcinoma; Head; Neck
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — temsirolimus

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Temsirolimus

SUMMARY:
This is an open-label, exploratory, biomarker study of intravenous temsirolimus given once weekly for 3 weeks to newly diagnosed, advanced stage head and neck cancer subjects prior to beginning their standard therapy for their specific disease. The primary objective of this study is to identify biomarkers of temsirolimus activity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with newly diagnosed, advanced stage, head and neck squamous cell carcinoma of the oral cavity, oral pharynx, hypopharynx or larynx.
* Subjects willing to undergo tumor biopsies.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Age >/= 18 years.

Exclusion Criteria:

* Subjects receiving anticoagulation therapy.
* Presence of unstable angina, recent myocardial infarction (within the previous 6 months), or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia.
* Prior cancer therapy (chemotherapy, hormonal therapy, radiotherapy, immunotherapy) or investigational agent for their head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Shreveport, Louisiana, United States